CLINICAL TRIAL: NCT06679907
Title: Cost-effectiveness Study Comparing Endovascular and Surgical Arteriovenous Fistula Creation for Haemodialysis in Patients with End-stage Renal Failure
Brief Title: Medico-economic Evaluation of the Creation of Arteriovenous Access for Hemodialysis Between Surgical Technique and Endovascular Technique in Patients with End-stage Renal Disease
Acronym: ENDOFAV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2023/49
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Endovascular Procedure; Hemodialysis
Keywords: Hemodialysis; arteriovenous; endovascular; restenosis; cost-effectiveness; health economic evaluation

STUDY DESIGN:
Intervention Model Description: Pragmatic, comparative, unblinded, randomized, controlled, prospective, parallel-arm multicenter superiority clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- WaveLinQ® device (Experimental): One of the two CE-marked devices used in the Endovascular AVF arm.
  Interventions: Device: WaveLinQ® device
- Ellipsys® device (Experimental): One of the two CE-marked devices used in the Endovascular AVF arm.
  Interventions: Device: Ellipsys® device
- Open surgery (Active Comparator)
  Interventions: Device: No device

INTERVENTIONS:
Device: WaveLinQ® device — The WaveLinQ® system employs a dual catheter technique to establish communication between deep arteries and veins, typically using a ulnar or radial artery and vein. This procedure necessitates fluoroscopic guidance to position the catheters correctly, a control angiogram, and potential embolization to enhance blood flow.
  Arms: WaveLinQ® device
Device: Ellipsys® device — The Ellipsys® system enables the entire AVF creation process to be conducted under ultrasound guidance without the need for fluoroscopy or contrast media. It uses a single needle to puncture the superficial vein, the perforator and the artery and potential balloon angioplasty to enhance blood flow.
  Arms: Ellipsys® device
Device: No device — Surgical AVF creation will involve a direct approach to the proximal radial, ulnar, or brachial artery to create a 4-6 mm longitudinal arteriotomy. An oblique incision will be made at the elbow crease. The cephalic, basilic, or perforating vein may be used for the side-to-end anastomosis. If a transposition is required due to adiposity, it will be performed either during the same procedure or at a later time through tunneling or lipectomy.
  Arms: Open surgery

SUMMARY:
This multicenter 1 :1 randomized controlled trial aims at comparing the cost-effectiveness of endovascular arteriovenous fistula (AVF) creation using Ellipsys® and WaveLinQ® devices with traditional surgical AVF creation for hemodialysis. The primary endpoint is the cost-utility ratio (cost per QALY gained), with an anticipated sample size of 252 patients. This study will provide critical insights into the viability and cost-effectiveness of endovascular techniques, potentially shaping future standards of care in hemodialysis access.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a global public health issue, affecting approximately 10% of the population.1,2 The number of patients starting renal replacement therapy has grown exponentially in recent years.3 Effective hemodialysis relies on a well-functioning vascular access (VA). The Kidney Disease Outcome Quality Initiative (KDOQI)4, the French Health Authority (HAS)5, and the European Society of Vascular and Endovascular Surgery (ESVS)6 recommend native arteriovenous fistulas (AVFs) as a primary option, referring to their lower morbidity, reduced mortality, and improved quality of life.7,8 An ideal AVF should allow cannulation with two needles, provide a blood flow of 300 to 600ml/min, resist infection and thrombosis, and have minimal adverse events.6 Between 2005 and 2007, 67-91% of patients in France used native AVFs.7 Data from the Dialysis Outcomes and Practice Patterns Study (DOPPS) showed that AVF maturation varies significantly by country, patient and center characteristics. In Japan, 84% of AVFs were created in the forearm, compared to 54% in EUR/ANZ (Belgium, France, Germany, Italy, Spain, Sweden, United Kingdom, Australia, and New Zealand), and 32% in the United States (US).9 Catheter-dependence following AVF creation remained high in EUR/ANZ and US patients, with nearly 70% still dependent 8 months after AVF creation. Failure to use AVFs within 6 months was associated to a 53% higher mortality rate in the following 6 months.9 A systematic review and meta-analysis of 318 studies10 reported that average AVF primary, assisted primary and secondary patency rates at one year were 64%, 73% and 79%, respectively. However, not all patent AVFs were suitable for dialysis: only 26% were mature at 6 months, and 21% were abandoned without ever being used.

Furthermore, up to 85% of AVFs require multiple re-interventions, including angioplasty, stenting, transposition, thrombectomy or thrombolysis within the first year.11-13 On average, up to 3.43 reinterventions per patient were required over the study duration, with higher rates for brachio-basilic accesses, contributing significantly to the overall cost of care.11-13 To improve outcomes, endovascular AVF creation techniques have been developed.14 These methods use radiofrequency or thermo-coagulation energy, guided by fluoroscopy and/or duplex ultrasound. Avoiding vessel dissection and mobilization, while minimizing trauma to the vascular wall and surrounding tissues, may help reduce the risk of intimal hyperplasia and AVF failure. This approach could lead to similar benefits as those demonstrated by surgical no-touch techniques.15 Preliminary results show a technical success rate of 97.5%, a 3-month maturation rate of 89.3%, a 1-year patency rate of 85.7%, and an average of 0.59 reinterventions per patient per year.16-19 As a results, data from the United States Renal Data System (USRDS) were compared to data from the Novel Endovascular Access Trial (NEAT) and both incident and prevalent patients with endoAVF required fewer interventions and had lower costs within the first year compared with matched patients with surgical AVFs.20 However, these devices are expensive (approximately €5,200 per patient) and the creation of an endovenous fistula is not yet listed in France's common classification of medical procedures (CCAM), making it ineligible for reimbursement by health insurance.21,22 In 2019, there were 15,653 hospitalizations in France for AVF creation and re-interventions to aid AVF maturation or restore patency in patients with end-stage renal disease. Although international studies suggest that endovascular AVF creation is effective,18,20,23 no French studies have yet replicated or confirmed these findings in the local context to support reimbursement claims. The 2018 ESVS guidelines also cite a lack of evidence on endovascular AVF creation.6 This protocol represents the first French medico-economic study to compare the two available endovascular AVF creation devices - Ellipsys® (Medtronic, Dublin, Ireland) and WaveLinQ® (BD, Bard, Franklin Lakes, New Jersey, United States of America) - with traditional open surgery. This randomized clinical trial aims to provide crucial data for healthcare decision-makers, potentially paving the way for the adoption of these devices in France, enhancing patient care, and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Age> 18 years
* On chronic dialysis, or due to start chronic dialysis within 3 to 6 months
* Patient eligible for the creation of a native surgical AVF at the elbow crease and an endovenous AVF according to the instructions for use of the manufacturers of the two devices used, namely:
* Target venous diameter for fistula creation > or = 3 mm
* Target arterial diameter for fistula creation > or = 2 mm
* Artery to vein distance < or = 1.5mm
* At least one superficial outflow vein with a diameter ≥ 2.5 mm connected via a proximal forearm perforating vein with the target site
* Patency of the radial and ulnar arteries confirmed by Doppler ultrasound
* Presence of a connecting perforator between the deep and superficial venous network, relatively straight anatomy
* Distance between proximal radial artery and perforator junction/radial vein < 1.5mm
* Patient having been clearly informed about the study and having agreed to participate and attend follow-up visits
* Patient affiliated or beneficiary of a social security scheme.

Exclusion Criteria:

* Known central venous stenosis > 50% on imaging or presence of an indwelling central venous catheter or pacemaker on the same side as the side of creation of the AVF
* Upper extremity arterial occlusive disease not amenable to endovascular or open repair
* Eligibility for a native distal AVF (radio or ulno-cephalic)
* New York Heart Association (NYHA) class III or IV heart failure
* Hypercoagulable state
* Estimated life expectancy <1 year
* Pregnantly or breastfeeding woman
* Known allergies to medical devices and medications used in the protocol
* Inability to collect consent
* Patient not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2030-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Cost-utility differential ratio (expressed as cost per Quality-Adjusted Life Year [QALY]) with endovascular AVF vs. open surgery | month 18
  This measure evaluates the cost-utility ratio by calculating the cost per QALY gained with the creation of an endovascular AVF using WaveLinQ® or Ellipsys® devices compared to an open surgical approach at 18 months. The assessment includes initial hospitalization costs via micro-costing and outpatient costs derived from the National Health Data System (SNDS) and evaluates utility using the EQ-5D-5L questionnaire.

SECONDARY OUTCOMES:
Evaluation of total cost of care for endovascular | Month 18
  This measure evaluates the total cost of care for endovascular AVF compared to surgical AVF creation at 18 and 36 months from the perspective of Mandatory Health Insurance.
Real costs of initial hospitalization for endovascular AVF vs. surgical AVF creation | Day 0
  This measure compares the real costs associated with the initial hospitalization for endovascular versus surgical AVF creation procedures.
Evaluation of total cost of care for surgical AVF creation | Month 18
  This measure evaluates the total cost of care for endovascular AVF compared to surgical AVF creation at 18 and 36 months from the perspective of Mandatory Health Insurance.
Evaluation of total cost of care for endovascular | Month 36
  This measure evaluates the total cost of care for endovascular AVF compared to surgical AVF creation at 18 and 36 months from the perspective of Mandatory Health Insurance.
Evaluation of total cost of care for surgical AVF creation | Month 36
  This measure evaluates the total cost of care for endovascular AVF compared to surgical AVF creation at 18 and 36 months from the perspective of Mandatory Health Insurance.
Evaluation of cost functional AVF without reintervention | Month 36
  This measure assesses the cost-effectiveness ratio as the cost per additional functional AVF without the need for reintervention at 36 months for WaveLinQ® or Ellipsys® devices compared to open surgery.
Evaluation of cost with adoption of endovascular AVF | 5 years
  Cost differences for health insurance over 5 years based on the adoption of endovascular techniques for AVF creation in patients requiring hemodialysis within 3-6 months or those already on dialysis in France. Data linkage between the clinical trial and the SNDS database will be performed through indirect matching using: age, postal code of residence, gender, date of hospital discharge, Diagnosis-Related Group Discharge Summary Code (GHM RSS), principal diagnosis of the stay, associated diagnoses, related diagnosis, stay number (NDA). Matching will enable continued follow-up without additional data collection, relying solely on SNIIRAM and PMSI data ensuring comprehensive tracking of AVF-related events across different care settings. Social determinants of health such as education, access to healthcare, housing stability, and socioeconomic status, will also be searched for to assess their po
Evaluation of frequency of reinterventions for vascular access | Month 36
  This measure calculates the frequency of reinterventions, including angioplasties, thrombectomies, AVF repairs, and new AVF creations, for each type of AVF creation. Data is derived from the French National Hospital Discharge Database (PMSI) and the French National Health Insurance Inter-Scheme Information System (SNIIRAM), with healthcare costs estimated from the SNDS.
Number of AVF creation success | Day 0
  This clinical endpoint measures the success rate of AVF creation. AVF creation success will be determined by the presence of a palpable "thrill" and/or confirmation of patency via immediate postoperative duplex scan.
Number of mature AVFs | Month 6
  This measure includes the proportion of AVFs that reach maturity and the time required for each AVF to mature, assessed at specific intervals. For dialysis patients, AVFs maturity will be defined as a vascular access allowing cannulation with two needles and providing adequate blood flow throughout hemodialysis. In pre-dialysis patients, maturity will be indicated by a pre-anastomotic humeral artery blood flow of at least 400 mL/min and an AVF diameter of at least 4 mm. AVF maturation time will be defined as the number of days between AVF creation and physiological maturation.
Number of mature AVFs | Month 12
  This measure includes the proportion of AVFs that reach maturity and the time required for each AVF to mature, assessed at specific intervals. For dialysis patients, AVFs maturity will be defined as a vascular access allowing cannulation with two needles and providing adequate blood flow throughout hemodialysis. In pre-dialysis patients, maturity will be indicated by a pre-anastomotic humeral artery blood flow of at least 400 mL/min and an AVF diameter of at least 4 mm. AVF maturation time will be defined as the number of days between AVF creation and physiological maturation.
Number of mature AVFs | Month 18
  This measure includes the proportion of AVFs that reach maturity and the time required for each AVF to mature, assessed at specific intervals. For dialysis patients, AVFs maturity will be defined as a vascular access allowing cannulation with two needles and providing adequate blood flow throughout hemodialysis. In pre-dialysis patients, maturity will be indicated by a pre-anastomotic humeral artery blood flow of at least 400 mL/min and an AVF diameter of at least 4 mm. AVF maturation time will be defined as the number of days between AVF creation and physiological maturation.
Evaluation of time to maturation | Month 6
  This measure includes the proportion of AVFs that reach maturity and the time required for each AVF to mature, assessed at specific intervals. For dialysis patients, AVFs maturity will be defined as a vascular access allowing cannulation with two needles and providing adequate blood flow throughout hemodialysis. In pre-dialysis patients, maturity will be indicated by a pre-anastomotic humeral artery blood flow of at least 400 mL/min and an AVF diameter of at least 4 mm. AVF maturation time will be defined as the number of days between AVF creation and physiological maturation.
Evaluation of time to maturation | Month 18
  This measure includes the proportion of AVFs that reach maturity and the time required for each AVF to mature, assessed at specific intervals. For dialysis patients, AVFs maturity will be defined as a vascular access allowing cannulation with two needles and providing adequate blood flow throughout hemodialysis. In pre-dialysis patients, maturity will be indicated by a pre-anastomotic humeral artery blood flow of at least 400 mL/min and an AVF diameter of at least 4 mm. AVF maturation time will be defined as the number of days between AVF creation and physiological maturation.
Evaluation of time to maturation | Month 12
  This measure includes the proportion of AVFs that reach maturity and the time required for each AVF to mature, assessed at specific intervals. For dialysis patients, AVFs maturity will be defined as a vascular access allowing cannulation with two needles and providing adequate blood flow throughout hemodialysis. In pre-dialysis patients, maturity will be indicated by a pre-anastomotic humeral artery blood flow of at least 400 mL/min and an AVF diameter of at least 4 mm. AVF maturation time will be defined as the number of days between AVF creation and physiological maturation.
Number of Functional AVFs | Month 6
  This measure evaluates the proportion of functional AVFs and assesses the recirculation rate, indicating access efficiency. AVFs functionality will be defined as a VA allowing successful cannulation with two needles over at least six hemodialysis sessions within 30 days, delivering satisfactory blood flow and achieving adequate dialysis (typically a minimum of 300 mL/min).
Number of Functional AVFs | Month 12
  This measure evaluates the proportion of functional AVFs and assesses the recirculation rate, indicating access efficiency. AVFs functionality will be defined as a VA allowing successful cannulation with two needles over at least six hemodialysis sessions within 30 days, delivering satisfactory blood flow and achieving adequate dialysis (typically a minimum of 300 mL/min).
Number of Functional AVFs | Month 18
  This measure evaluates the proportion of functional AVFs and assesses the recirculation rate, indicating access efficiency. AVFs functionality will be defined as a VA allowing successful cannulation with two needles over at least six hemodialysis sessions within 30 days, delivering satisfactory blood flow and achieving adequate dialysis (typically a minimum of 300 mL/min).
Number of recirculation | Month 6
  This measure evaluates the proportion of functional AVFs and assesses the recirculation rate, indicating access efficiency. The recirculation rate will refer to the percentage of dialyzed blood that re-enters the systemic circulation without complete clearance.
Number of recirculation | Month 12
  This measure evaluates the proportion of functional AVFs and assesses the recirculation rate, indicating access efficiency. The recirculation rate will refer to the percentage of dialyzed blood that re-enters the systemic circulation without complete clearance.
Number of recirculation | Month 18
  This measure evaluates the proportion of functional AVFs and assesses the recirculation rate, indicating access efficiency. The recirculation rate will refer to the percentage of dialyzed blood that re-enters the systemic circulation without complete clearance.
Number of days hospitalised for AVF creation | Day 15
  This measure records the average length of stay, in days, for initial hospitalization associated with AVF creation.
Number of adverse events related to vascular access | Day 1
  his measure monitors complications arising from vascular access, including limb ischemia (steal syndrome), monomelic ischemic neuropathy, high-flow conditions (blood flow > 1500 mL/min with cardiac consequences), aneurysms, hemorrhages, skin necrosis, infections, thrombosis, and AVF abandonment, with ischemia severity classified into four stages ranging from mild coldness and numbness (stage 1) to tissue loss affecting the extremities (stage 4)
Number of adverse events related to vascular access | Month 1
  his measure monitors complications arising from vascular access, including limb ischemia (steal syndrome), monomelic ischemic neuropathy, high-flow conditions (blood flow > 1500 mL/min with cardiac consequences), aneurysms, hemorrhages, skin necrosis, infections, thrombosis, and AVF abandonment, with ischemia severity classified into four stages ranging from mild coldness and numbness (stage 1) to tissue loss affecting the extremities (stage 4)
Number of adverse events related to vascular access | Month 6
  his measure monitors complications arising from vascular access, including limb ischemia (steal syndrome), monomelic ischemic neuropathy, high-flow conditions (blood flow > 1500 mL/min with cardiac consequences), aneurysms, hemorrhages, skin necrosis, infections, thrombosis, and AVF abandonment, with ischemia severity classified into four stages ranging from mild coldness and numbness (stage 1) to tissue loss affecting the extremities (stage 4)
Number of adverse events related to vascular access | Month 12
  his measure monitors complications arising from vascular access, including limb ischemia (steal syndrome), monomelic ischemic neuropathy, high-flow conditions (blood flow > 1500 mL/min with cardiac consequences), aneurysms, hemorrhages, skin necrosis, infections, thrombosis, and AVF abandonment, with ischemia severity classified into four stages ranging from mild coldness and numbness (stage 1) to tissue loss affecting the extremities (stage 4)
Number of adverse events related to vascular access | Month 18
  his measure monitors complications arising from vascular access, including limb ischemia (steal syndrome), monomelic ischemic neuropathy, high-flow conditions (blood flow > 1500 mL/min with cardiac consequences), aneurysms, hemorrhages, skin necrosis, infections, thrombosis, and AVF abandonment, with ischemia severity classified into four stages ranging from mild coldness and numbness (stage 1) to tissue loss affecting the extremities (stage 4)
Number of serious adverse events related to AVF device | Day 0
  This measure tracks serious adverse events directly related to the AVF device.
Number of serious adverse events related to AVF device | Month 1
  This measure tracks serious adverse events directly related to the AVF device.
Number of serious adverse events related to AVF device | Month 6
  This measure tracks serious adverse events directly related to the AVF device.
Number of serious adverse events related to AVF device | Month 12
  This measure tracks serious adverse events directly related to the AVF device.
Number of serious adverse events related to AVF device | Month 18
  This measure tracks serious adverse events directly related to the AVF device.
Number of serious adverse events related to AVF device | Month 36
  This measure tracks serious adverse events directly related to the AVF device.
Number of Reinterventions related to AVF device | Day 0
  This measure tracks early reinterventions (within 1 month) and late reinterventions (after 1 month) such as angioplasties, thrombectomies, AVF repairs, and new AVF creations.
Number of Reinterventions related to AVF device | Month 1
  This measure tracks early reinterventions (within 1 month) and late reinterventions (after 1 month) such as angioplasties, thrombectomies, AVF repairs, and new AVF creations.
Number of Reinterventions related to AVF device | Month 6
  This measure tracks early reinterventions (within 1 month) and late reinterventions (after 1 month) such as angioplasties, thrombectomies, AVF repairs, and new AVF creations.
Number of Reinterventions related to AVF device | Month 12
  This measure tracks early reinterventions (within 1 month) and late reinterventions (after 1 month) such as angioplasties, thrombectomies, AVF repairs, and new AVF creations.
Number of Reinterventions related to AVF device | Month 18
  This measure tracks early reinterventions (within 1 month) and late reinterventions (after 1 month) such as angioplasties, thrombectomies, AVF repairs, and new AVF creations.
Number of Reinterventions related to AVF device | Month 36
  This measure tracks early reinterventions (within 1 month) and late reinterventions (after 1 month) such as angioplasties, thrombectomies, AVF repairs, and new AVF creations.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine - Centre Aquitain des pathologies vasculaire, Bordeaux
  - AP-HP Centre Hospitalier Universitaire d'Ambroise Paré, Boulogne-Billancourt
  - Clinique du parc, Castelnau-le-Lez
  - Centre Hospitalier Universitaire de Dijon - Hôpital le Bocage, Dijon
  - Centre Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital privé Jean Mermoz, Lyon
  - Centre Hospitalier St Joseph - St Luc, Lyon
  - Centre Hospitalier Universitaire de Nice - Hôpital Pasteur 1, Nice
  - Groupe Hospitalier Paris St Joseph - Centre Hospitalier Chartres, Paris
  - Centre Hospitalier Universitaire de Nantes - Hôpital Nord Laennec, Saint-Herblain

IPD SHARING:
Plan to Share IPD: Yes
The data is available from Pr Eric DUCASSE . An email can be sent to her so that she can contact the data manager and owner, the Bordeaux University Hospital. The data can be made available after contractual agreement.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Jones RG, Morgan RA. A Review of the Current Status of Percutaneous Endovascular Arteriovenous Fistula Creation for Haemodialysis Access. Cardiovasc Intervent Radiol. 2019 Jan;42(1):1-9. doi: 10.1007/s00270-018-2037-6. Epub 2018 Jul 20. PMID 30030582
- [Background] Arnold RJG, Han Y, Balakrishnan R, Layton A, Lok CE, Glickman M, Rajan DK. Comparison between Surgical and Endovascular Hemodialysis Arteriovenous Fistula Interventions and Associated Costs. J Vasc Interv Radiol. 2018 Nov;29(11):1558-1566.e2. doi: 10.1016/j.jvir.2018.05.014. Epub 2018 Oct 5. PMID 30293731
- [Background] Shahverdyan R, Beathard G, Mushtaq N, Litchfield TF, Nelson PR, Jennings WC. Comparison of Outcomes of Percutaneous Arteriovenous Fistulae Creation by Ellipsys and WavelinQ Devices. J Vasc Interv Radiol. 2020 Sep;31(9):1365-1372. doi: 10.1016/j.jvir.2020.06.008. Epub 2020 Aug 11. PMID 32792280
- [Background] Mallios A, Bourquelot P, Franco G, Hebibi H, Fonkoua H, Allouache M, Costanzo A, de Blic R, Harika G, Boura B, Jennings WC. Midterm results of percutaneous arteriovenous fistula creation with the Ellipsys Vascular Access System, technical recommendations, and an algorithm for maintenance. J Vasc Surg. 2020 Dec;72(6):2097-2106. doi: 10.1016/j.jvs.2020.02.048. Epub 2020 Apr 8. PMID 32276012
- [Background] Hull J, Deitrick J, Groome K. Maturation for Hemodialysis in the Ellipsys Post-Market Registry. J Vasc Interv Radiol. 2020 Sep;31(9):1373-1381. doi: 10.1016/j.jvir.2020.03.001. Epub 2020 Aug 14. PMID 32800660
- [Background] Mallios A, Jennings WC, Boura B, Costanzo A, Bourquelot P, Combes M. Early results of percutaneous arteriovenous fistula creation with the Ellipsys Vascular Access System. J Vasc Surg. 2018 Oct;68(4):1150-1156. doi: 10.1016/j.jvs.2018.01.036. Epub 2018 Apr 19. PMID 29680297
- [Background] Bhojani MF, Malik J, Mumtaz A, Sophie Z, Waseem S. Beyond Conventional: A Systematic Review of Non-Conventional Techniques for Radio-Cephalic Arteriovenous Fistula. Ann Vasc Surg. 2025 Jan;110(Pt B):306-316. doi: 10.1016/j.avsg.2024.07.091. Epub 2024 Aug 7. PMID 39096957
- [Background] Rajan DK, Lok CE. Promises for the future: minimally invasive fistula creation. J Vasc Access. 2015;16 Suppl 9:S40-1. doi: 10.5301/jva.5000351. Epub 2015 Mar 8. PMID 25751549
- [Background] Palmes D, Kebschull L, Schaefer RM, Pelster F, Konner K. Perforating vein fistula is superior to forearm fistula in elderly haemodialysis patients with diabetes and arterial hypertension. Nephrol Dial Transplant. 2011 Oct;26(10):3309-14. doi: 10.1093/ndt/gfr004. Epub 2011 Feb 16. PMID 21325347
- [Background] Koksoy C, Demirci RK, Balci D, Solak T, Kose SK. Brachiobasilic versus brachiocephalic arteriovenous fistula: a prospective randomized study. J Vasc Surg. 2009 Jan;49(1):171-177.e5. doi: 10.1016/j.jvs.2008.08.002. Epub 2008 Oct 22. PMID 18945577
- [Background] Woo K, Farber A, Doros G, Killeen K, Kohanzadeh S. Evaluation of the efficacy of the transposed upper arm arteriovenous fistula: a single institutional review of 190 basilic and cephalic vein transposition procedures. J Vasc Surg. 2007 Jul;46(1):94-99; discussion 100. doi: 10.1016/j.jvs.2007.02.057. Epub 2007 Jun 1. PMID 17543490
- [Background] Bylsma LC, Gage SM, Reichert H, Dahl SLM, Lawson JH. Arteriovenous Fistulae for Haemodialysis: A Systematic Review and Meta-analysis of Efficacy and Safety Outcomes. Eur J Vasc Endovasc Surg. 2017 Oct;54(4):513-522. doi: 10.1016/j.ejvs.2017.06.024. Epub 2017 Aug 23. PMID 28843984
- [Background] Pisoni RL, Zepel L, Zhao J, Burke S, Lok CE, Woodside KJ, Wasse H, Kawanishi H, Schaubel DE, Zee J, Robinson BM. International Comparisons of Native Arteriovenous Fistula Patency and Time to Becoming Catheter-Free: Findings From the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2021 Feb;77(2):245-254. doi: 10.1053/j.ajkd.2020.06.020. Epub 2020 Sep 21. PMID 32971192
- [Background] Ravani P, Palmer SC, Oliver MJ, Quinn RR, MacRae JM, Tai DJ, Pannu NI, Thomas C, Hemmelgarn BR, Craig JC, Manns B, Tonelli M, Strippoli GF, James MT. Associations between hemodialysis access type and clinical outcomes: a systematic review. J Am Soc Nephrol. 2013 Feb;24(3):465-73. doi: 10.1681/ASN.2012070643. Epub 2013 Feb 21. PMID 23431075
- [Background] Ethier J, Mendelssohn DC, Elder SJ, Hasegawa T, Akizawa T, Akiba T, Canaud BJ, Pisoni RL. Vascular access use and outcomes: an international perspective from the Dialysis Outcomes and Practice Patterns Study. Nephrol Dial Transplant. 2008 Oct;23(10):3219-26. doi: 10.1093/ndt/gfn261. Epub 2008 May 29. PMID 18511606
- [Background] Schmidli J, Widmer MK, Basile C, de Donato G, Gallieni M, Gibbons CP, Haage P, Hamilton G, Hedin U, Kamper L, Lazarides MK, Lindsey B, Mestres G, Pegoraro M, Roy J, Setacci C, Shemesh D, Tordoir JHM, van Loon M, Esvs Guidelines Committee, Kolh P, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Lindholt J, Naylor R, Vega de Ceniga M, Vermassen F, Verzini F, Esvs Guidelines Reviewers, Mohaupt M, Ricco JB, Roca-Tey R. Editor's Choice - Vascular Access: 2018 Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Jun;55(6):757-818. doi: 10.1016/j.ejvs.2018.02.001. Epub 2018 May 2. No abstract available. PMID 29730128
- [Background] Erratum Regarding "KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update" (Am J Kidney Dis. 2020;75[4][suppl 2]:S1-S164). Am J Kidney Dis. 2021 Apr;77(4):551. doi: 10.1053/j.ajkd.2021.02.002. No abstract available. PMID 33752805
- [Background] Port FK. End-stage renal disease: magnitude of the problem, prognosis of future trends and possible solutions. Kidney Int Suppl. 1995 Aug;50:S3-6. PMID 8544432
- [Background] Wetzels JF, Kiemeney LA, Swinkels DW, Willems HL, den Heijer M. Age- and gender-specific reference values of estimated GFR in Caucasians: the Nijmegen Biomedical Study. Kidney Int. 2007 Sep;72(5):632-7. doi: 10.1038/sj.ki.5002374. Epub 2007 Jun 13. PMID 17568781
- [Background] Coresh J, Astor BC, Greene T, Eknoyan G, Levey AS. Prevalence of chronic kidney disease and decreased kidney function in the adult US population: Third National Health and Nutrition Examination Survey. Am J Kidney Dis. 2003 Jan;41(1):1-12. doi: 10.1053/ajkd.2003.50007. PMID 12500213